CLINICAL TRIAL: NCT01349907
Title: A 50-Week Open-Label, Flexible-Dose Trial of Asenapine Extension Treatment to P06107 in Pediatric Subjects With Acute Manic or Mixed Episodes Associated With Bipolar I Disorder
Brief Title: Extension Study of Asenapine [P06107 (NCT01244815)] for Pediatric Bipolar Disorder (P05898)
Acronym: ADDRESS-98
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05898; MK-8274-022 (Other: Merck Protocol Number)
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2022-02

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — asenapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Asenapine/Asenapine (Experimental): Participants treated with asenapine in base trial P06107, were first treated with open-label flavored asenapine 2.5 mg twice per day (BID), then up-titrated to 5 mg BID at day 4, then up-titrated to 10 mg BID at Day 7. After Day 7, flexible dosing of asenapine was continued for up to 50 weeks.
  Interventions: Drug: Asenapine; Drug: Rescue medication
- Placebo/Asenapine (Experimental): Participants treated with placebo in base trial P06107, were first treated with open-label flavored asenapine 2.5 mg BID, then up-titrated to 5 mg BID at day 4, then up-titrated to 10 mg BID at Day 7. After Day 7, flexible dosing of asenapine was continued for up to 50 weeks.
  Interventions: Drug: Asenapine; Drug: Rescue medication

INTERVENTIONS:
Drug: Asenapine — One flavored asenapine sublingual tablet (containing either 2.5, 5 or 10 mg asenapine) twice daily (BID), starting at 2.5 mg on Day 1 for three consecutive days. Normally on Day 4, the dose will increase to 5 mg BID beginning with the evening dose. Normally on Day 7, the dose will increase to 10 mg BID beginning with the evening dose. The dose may be up-titrated earlier than Days 4 and 7 at the investigator's discretion. Beginning on Day 8 (or after at least 1 day on 10 mg BID), asenapine dosing will be flexible (2.5, 5, or 10 mg BID) until up to Week 50.
  Other Names: SCH 900274, ORG 5222
Drug: Rescue medication — For participants whose symptoms worsen or are not adequately controlled on assigned treatment, rescue medication may be administered during the trial in the following circumstances. For the control of agitation, anxiety, insomnia, restlessness, or akathisia and extrapyramidal symptoms (EPS) some benzodiazepines (i.e., lorazepam [up to 4 mg/day] or an equivalent dose of short-acting benzodiazepines) and EPS medications (i.e., anticholinergics) are allowed. Benadryl (diphenhydramine) and beta blockers are also permitted, provided that they are not taken within 8 hours of efficacy assessments.

SUMMARY:
This study will investigate the safety and tolerability of a flexible dosing regimen of asenapine for the long-term treatment of manic or mixed episodes associated with bipolar disorder I in children and adolescents who completed study P06107.

ELIGIBILITY:
Inclusion Criteria:

* Completed study P06107 and demonstrated acceptable degree of compliance with medication, visits and other study requirements
* Must be male or a female who is not of childbearing potential and is not sexually active or is using a medically accepted method of contraception; or female who is not pregnant, or not lactating.
* Must have a caregiver or responsible person living with the participant who agrees to provide support to ensure compliance with treatment, visits, and protocol procedures

Exclusion Criteria:

* Positive pregnancy test or intention to become pregnant during the study
* At imminent risk of self-harm or harm to others
* Under involuntary inpatient commitment
* Known serological evidence of human immunodeficiency virus (HIV) antibody

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 322 (Actual)
Dates: Start 2011-06-16 (Actual); Primary Completion 2014-09-05 (Actual); Study Completion 2014-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Findling RL, Landbloom RL, Szegedi A, Koppenhaver J, Braat S, Zhu Q, Mackle M, Chang K, Mathews M. Asenapine for the Acute Treatment of Pediatric Manic or Mixed Episode of Bipolar I Disorder. J Am Acad Child Adolesc Psychiatry. 2015 Dec;54(12):1032-41. doi: 10.1016/j.jaac.2015.09.007. Epub 2015 Oct 24. PMID 26598478
- [Derived] Findling RL, Landbloom RL, Mackle M, Wu X, Snow-Adami L, Chang K, Durgam S. Long-term Safety of Asenapine in Pediatric Patients Diagnosed With Bipolar I Disorder: A 50-Week Open-Label, Flexible-Dose Trial. Paediatr Drugs. 2016 Oct;18(5):367-78. doi: 10.1007/s40272-016-0184-2. PMID 27461426

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a diagnosis of bipolar I disorder who completed the 3-week base trial P06107 (NCT01224485).
Groups:
- Asenapine/Asenapine: Participants treated with asenapine in base trial P06107, were first treated with open-label flavored asenapine 2.5 mg twice daily (BID), then up-titrated to 5 mg BID at day 4, then up-titrated to 10 mg BID at Day 7. After Day 7, flexible dosing of asenapine was continued for up to 50 weeks.
Period: Overall Study
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Started | 241 (Enrolled and Treated) | 81 (Enrolled and Treated)
Completed | 102 | 38
Not Completed | 139 | 43
Not completed — Adverse Event | 37 | 11
Not completed — Treatment failure | 13 | 4
Not completed — Lost to Follow-up | 25 | 6
Not completed — Withdrawal by Subject | 30 | 8
Not completed — Protocol Violation | 33 | 13
Not completed — Administrative | 1 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of trial medication, and were 17 years old or younger. One 18 year old participant from the Placebo/Asenapine group, was excluded due to being overage.
Groups:
- Asenapine/Asenapine: Participants treated with asenapine in base trial P06107 were first treated with open-label flavored asenapine 2.5 mg BID, then up-titrated to 5 mg BID at day 4, then up-titrated to 10 mg BID at Day 7. After Day 7, flexible dosing of asenapine was continued for up to 50 weeks.
- Total: Total of all reporting groups
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine | Total
Number analyzed (Participants) | 241 | 80 | 321
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.8 (2.0) | 13.7 (2.0) | 13.8 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 47 | 160
  Male | 128 | 33 | 161

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Clinical or Laboratory Adverse Events
Description: A clinical or laboratory adverse event is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product.
Time Frame: Baseline (Day 1) to 30 days after the last dose of study drug (up to approximately 54 weeks)
Population: Participants who received at least one dose of trial medication, and were 17 years old or younger. One treated participant from the Placebo/Asenapine group, who was 18 years old, was excluded from this analysis.
Measure: Number; unit: Participants
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Number analyzed (Participants) | 241 | 80
Participants | 197 | 74

2. Secondary Outcome: Change From Baseline in Young Mania Rating Scale (Y-MRS) Total Score
Description: The Y-MRS assesses the severity of manic episodes by assigning a severity rating to each of 11 items (Elevated mood, Increased motor activity-energy, Sexual interest, Sleep, Irritability, Speech, Language-thought disorder, Thought content, Disruptive-aggressive behavior, Appearance, Insight). Seven of the 11 items are rated on a scale of 0-4, and 4 of the items are rated on a scale of 0-8. The Y-MRS total score, observed cases (OC), the assessment closest to the scheduled assessment day within the allowed window, is the sum of the ratings for the 11 individual items, and can range from 0-60, with higher scores indicating greater severity of symptoms. Improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline, Day 182 and Day 350
Population: Participants 17 years old or younger, who have taken at least one dose of trial medication, and have a baseline, and at least one post-baseline Y-MRS assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Number analyzed (Participants) | 227 | 72
Score on a scale
  Day 182 (n=112, 37) | -4.9 (7.8) | -13.0 (8.3)
  Day 350 (n=45, 20) | -6.5 (10.5) | -15.2 (5.8)

3. Secondary Outcome: Percentage of Participants Who Were Y-MRS Total Score Remitters (Y-MRS ≤12)
Description: The Y-MRS is an 11-item clinician-rated instrument for assessing the severity of manic episodes. The Y-MRS total score, OC for each participant is the sum of the ratings for the 11 individual items, and can range from 0-60, with higher scores indicating greater severity of symptoms. A remitter is a participant with a Y-MRS total score of 12 or lower.
Time Frame: Up to Day 350
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Number analyzed (Participants) | 227 | 72
Percentage of participants
  Day 182 (n= 112, 37) | 63.4 | 83.8
  Day 350 (n = 45, 20) | 75.6 | 90.0

4. Secondary Outcome: Percentage of Participants Who Were Y-MRS Total Score Responders
Description: The Y-MRS is an 11-item clinician-rated instrument for assessing the severity of manic episodes. The Y-MRS total score, OC for each participant is the sum of the ratings for the 11 individual items, and can range from 0-60, with higher scores indicating greater severity of symptoms. A Y-MRS responder experiences a 50% or more decrease from baseline in Y-MRS total score.
Time Frame: Up to Day 350
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Number analyzed (Participants) | 227 | 72
Percentage of participants
  Day 182 (n= 111, 37) | 37.8 | 64.9
  Day 350 (n=43, 20) | 53.5 | 80.0

5. Secondary Outcome: Time to First Total Y-MRS 50% Response
Description: The Y-MRS is an 11-item clinician-rated instrument for assessing the severity of manic episodes. The Y-MRS total score, OC for each participant is the sum of the ratings for the 11 individual items, ranging from 0-60, with higher scores indicating more severe symptoms. The time to 50% response is the number of days on treatment to achieve a 50% decrease from baseline in Y-MRS total score.
Time Frame: Up to Day 350
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Number analyzed (Participants) | 227 | 72
Days | 15.0 [14.0 to 21.0] | 49.0 [44.0 to 50.0]

6. Secondary Outcome: Time to Failure to Maintain Response in Y-MRS Total Score
Description: The Y-MRS is an 11-item clinician-rated instrument for assessing the severity of manic episodes. The Y-MRS total score, OC for each participant is the sum of the ratings for the 11 individual items, ranging from 0-60, with higher scores indicating more severe symptoms. The time to failure is the number of days from first achieving a 50% or more decrease from baseline in Y-MRS total score to the first subsequent day of a less than 50% decrease from baseline in Y-MRS total score.
Time Frame: Up to Day 350
Population: Participants 17 years old or younger, who have taken at least one dose of trial medication, and have a baseline, and at least one post-baseline Y-MRS assessment. Restricted to participants who were total Y-MRS 50% responders in base trial P06107.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Number analyzed (Participants) | 120 | 21
Days | NA [268.0 to NA] — NA = Not achieved after 362 days of follow-up | 194.0 [78.0 to NA] — NA = Not achieved after 362 days of follow-up

7. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale for Assessing Overall Bipolar Illness (CGI-BP Overall)
Description: The CGI-BP overall is a single value score OC for assessing overall bipolar illness, recorded on a 7-point scale ranging from 1 for normal/not ill, to 7 for very severely ill. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline, Day 182 and Day 350
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Number analyzed (Participants) | 227 | 72
Score on a scale
  Day 182 (n=113, 37) | -0.9 (1.0) | -1.8 (1.1)
  Day 350 (n=46, 20) | -1.2 (1.3) | -2.4 (1.2)

8. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale for Assessing Depression (CGI-BP Depression)
Description: The CGI-BP depression is a single value score OC for assessing depression, recorded on a 7-point scale ranging from 1 for normal/not ill, to 7 for very severely ill. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline, Day 182 and Day 350
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Number analyzed (Participants) | 227 | 72
Score on a scale
  Day 182 (n=113, 37) | -0.5 (0.9) | -0.8 (1.2)
  Day 350 (n=46, 20) | -0.4 (1.0) | -1.2 (1.3)

9. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale for Assessing Mania (CGI-BP Mania)
Description: The CGI-BP mania is a single value score OC for assessing mania, recorded on a 7-point scale ranging from 1 for normal/not ill, to 7 for very severely ill. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline, Day 182 and Day 350
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Number analyzed (Participants) | 227 | 72
Score on a scale
  Day 182 (n=113, 37) | -1.0 (1.0) | -1.9 (1.1)
  Day 350 (n=46, 20) | -1.2 (1.3) | -2.3 (1.2)

10. Secondary Outcome: Change From Baseline in Children's Depression Rating Scale, Revised (CDRS-R) Total Score
Description: The CDRS-R is a 17-item clinician-rated instrument for assessing the presence and severity of depressive symptoms in children. Fourteen of the 17 items are rated on a scale of 1-7, and 3 of the items are rated on a scale of 1-5, with higher scores indicating greater severity of symptoms. The CDRS-R total score, OC for each participant is the sum of the ratings for the 17 individual items, and can range from 17-113, with higher scores indicating greater severity of symptoms. Improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline, Day 182 and Day 350
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Number analyzed (Participants) | 227 | 72
Score on a scale
  Day 182 (n=112, 37) | -1.4 (6.4) | -5.4 (7.5)
  Day 350 (n=44, 20) | -1.1 (5.5) | -4.3 (6.6)

11. Secondary Outcome: Percentage of CDRS-R Responders
Description: The CDRS-R is a 17-item clinician-rated instrument for assessing the presence and severity of depressive symptoms in children. The CDRS-R total score, OC for each participant is the sum of the ratings for the 17 individual items, and can range from 17-113, with higher scores indicating greater severity of symptoms. A CDRS-R responder experiences a 50% or more decrease from baseline in CDRS-R total score.
Time Frame: Up to Day 350
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Number analyzed (Participants) | 227 | 72
Percentage of participants
  Day 182 (n=111, 37) | 36.0 | 56.8
  Day 350 (n=43, 20) | 32.6 | 65.0

12. Secondary Outcome: Percentage of Participants With Emergent Depression Based on CDRS-R
Description: The CDRS-R is a 17-item clinician-rated instrument for assessing the presence and severity of depressive symptoms in children. The CDRS-R total score, OC for each participant is the sum of the ratings for the 17 individual items, and can range from 17-113, with higher scores indicating greater severity of symptoms. Participants with a CDRS-R score of 40 or greater (whose baseline CDRS-R is less than 40) exhibit emergent depression, which is a strong indicator of the presence or potential for a major depressive disorder.
Time Frame: Up to Day 350
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Number analyzed (Participants) | 227 | 72
Percentage of participants
  Day 182 (n=112, 37) | 2.7 | 0.0
  Day 350 (n=44, 20) | 2.3 | 5.0

13. Secondary Outcome: Change From Baseline in Children's Global Assessment Scale (CGAS)
Description: CGAS is a scale with a possible range of 1 to 100, measuring psychological, social, and school functioning in children. Minimum scores, OC range from 1-10, representing the need for constant supervision (worse result) to maximum scores of 91-100, representing superior functioning (better result). An improvement in function is represented by a change from baseline value that is positive.
Time Frame: Baseline, Day 182 and Day 350
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Number analyzed (Participants) | 227 | 72
Score on a scale
  Day 182 (n=114, 37) | 9.7 (10.1) | 17.4 (9.9)
  Day 350 (n=46, 20) | 13.1 (13.6) | 22.5 (8.0)

14. Secondary Outcome: Percentage of Participants With a CGAS Score of Equal or Greater Than 70
Description: CGAS is a scale with a possible range of 1 to 100, measuring psychological, social, and school functioning in children. Minimum scores, OC range from 1-10, representing the need for constant supervision (worse result) to maximum scores of 91-100, representing superior functioning (better result). The percentage of participants with a score of 70 or greater, representing normal to superior social functioning, is shown.
Time Frame: Up to Day 350
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Number analyzed (Participants) | 227 | 72
Percentage of participants
  Day 182 (n=114, 37) | 55.3 | 73.0
  Day 350 (n=46, 20) | 73.9 | 85.0

15. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Enjoyment and Satisfaction Questionnaires (PQ-LES-Q) Total Score
Description: PQ-LES-Q is a questionnaire to assess quality of life enjoyment and satisfaction in children and adolescents. The participant rates 15 items reflecting quality of life from the previous week on a scale of 1=very poor to 5=very good. Items 1-14 assess specific areas (e.g., health, mood or feelings); item 15 is a global assessment of overall quality of life. The PQ-LES-Q total score for each participant, OC is the sum of the rating assigned to each of the first 14 items, and ranges from 14 to 70, with a higher score indicating better quality of life. An improvement in quality of life is represented by change from baseline values that are positive.
Time Frame: Baseline, Day 182 and Day 350
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Number analyzed (Participants) | 227 | 72
Score on a scale
  Day 182 (n=111, 36) | 1.0 (7.1) | 4.4 (8.3)
  Day 350 (n=45, 20) | 0.5 (7.3) | 3.4 (10.9)

16. Secondary Outcome: Change From Baseline in PQ-LES-Q Overall Score
Description: PQ-LES-Q is a questionnaire to assess quality of life enjoyment and satisfaction in children and adolescents. The participant rates 15 items reflecting quality of life from the previous week. Item 15, the PQ-LES-Q overall score, observed OC, is a global assessment of overall quality of life, and ranges from 1 to 5, with a higher score indicating better quality of life. An improvement in quality of life is represented by change from baseline values that are positive.
Time Frame: Baseline, Day 182 and Day 350
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Number analyzed (Participants) | 227 | 72
Score on a scale
  Day 182 (n=111, 36) | 0.1 (0.8) | 0.3 (0.8)
  Day 350 (n=45, 20) | 0.4 (1.0) | 0.3 (0.9)

ADVERSE EVENTS:
Time Frame: 30 days after the last dose of study drug (up to approximately 54 weeks).
Description: All enrolled and treated participants
Arm/Group | Asenapine/Asenapine | Placebo/Asenapine
Serious Adverse Events (participants affected / at risk) | 17/241 | 6/81
Other Adverse Events (participants affected / at risk) | 135/241 | 65/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine/Asenapine (N=241) | Placebo/Asenapine (N=81)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (2)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 2 (2) | 1 (2)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 2 (3) | 2 (2)
Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Disturbance in social behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Exhibitionism (Psychiatric disorders) | 1 (1) | 0 (0)
Impulsive behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Self-injurious ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 7 (8) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine/Asenapine (N=241) | Placebo/Asenapine (N=81)
Abdominal pain upper (Gastrointestinal disorders) | 10 (15) | 6 (6)
Hypoaesthesia oral (Gastrointestinal disorders) | 2 (2) | 11 (11)
Nausea (Gastrointestinal disorders) | 15 (17) | 9 (9)
Paraesthesia oral (Gastrointestinal disorders) | 3 (3) | 8 (10)
Vomiting (Gastrointestinal disorders) | 16 (18) | 4 (4)
Fatigue (General disorders) | 15 (17) | 6 (7)
Gastroenteritis viral (Infections and infestations) | 4 (4) | 5 (5)
Weight increased (Investigations) | 42 (43) | 16 (16)
Increased appetite (Metabolism and nutrition disorders) | 16 (18) | 6 (6)
Dizziness (Nervous system disorders) | 5 (6) | 8 (10)
Dysgeusia (Nervous system disorders) | 4 (4) | 5 (5)
Headache (Nervous system disorders) | 21 (30) | 11 (21)
Sedation (Nervous system disorders) | 23 (29) | 19 (27)
Somnolence (Nervous system disorders) | 44 (50) | 29 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication or manuscript shall contain any trade secret information of the sponsor or any proprietary or confidential information of the sponsor, and shall be confined to new discoveries and interpretations of scientific fact.